CLINICAL TRIAL: NCT03326245
Title: Dopaminergic Modulation of Brain Activation Using Simultaneous PET/Pharmacological MRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 170178; 17-AA-0178
Record Dates: First submitted 2017-10-28; First posted 2017-10-31 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-10-27

CONDITIONS: Normal Physiology
Keywords: Pharmacological MRI; C-11 Raclopride; PET Imaging; Neuropsychological Testing
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Oral methylphenidate followed by intravenous placebo (Active Comparator): Healthy participants receive methylphenidate 60mg orally given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous placebo (3ml saline) given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection. Participants were subsequently randomized across study arms B and C in different study days with at least 48 hours between visits.
  Interventions: Drug: Methylphenidate Pill; Drug: Intravenous Placebo
- Arm B: Oral placebo followed by intravenous methylphenidate (Active Comparator): Healthy participants receive oral placebo given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous methylphenidate 0.25 mg/kg in 3ml sterile water given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection. Participants were subsequently randomized across study arms A and C in different study days with at least 48 hours between visits.
  Interventions: Drug: Oral Placebo; Drug: Intravenous methylphenidate
- Arm C: Oral placebo followed by intravenous placebo (Placebo Comparator): Healthy participants receive oral placebo given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous placebo (3ml saline) given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection. Participants were subsequently randomized across study arms A and B in different study days with at least 48 hours between visits.
  Interventions: Drug: Oral Placebo; Drug: Intravenous Placebo

INTERVENTIONS:
Drug: Methylphenidate Pill — Oral methylphenidate (60 mg) given 30 minutes prior to bolus [11C]raclopride
  Other Names: Ritalin
  Arms: Arm A: Oral methylphenidate followed by intravenous placebo
Drug: Oral Placebo — Oral PL will be given 30 minutes prior to bolus [11C]raclopride injection
  Arms: Arm B: Oral placebo followed by intravenous methylphenidate; Arm C: Oral placebo followed by intravenous placebo
Drug: Intravenous Placebo — Intravenous Placebo given 30 minutes post bolus injection of [11C]raclopride.
  Arms: Arm A: Oral methylphenidate followed by intravenous placebo; Arm C: Oral placebo followed by intravenous placebo
Drug: Intravenous methylphenidate — Intravenous methylphenidate 0.25 mg/kg in 3ml sterile saline given 30 minutes post bolus injection of [11C]raclopride.
  Arms: Arm B: Oral placebo followed by intravenous methylphenidate

SUMMARY:
Background:

Dopamine (DA) is a chemical signal in the brain linked to learning, memory, and habits. Stimulant drugs like methylphenidate can increase DA in the brain. Researchers want to measure DA with and without this drug. They want to learn how methylphenidate and brain dopamine affect body responses, mood, and thinking.

Objective:

To better understand the role of dopamine in the brain and the effects of methylphenidate.

Eligibility:

Adults ages 18-55 who have used alcohol or stimulant drugs but have no drug dependence.

Design:

Participants will be screened with:

* Physical exam
* Question about medical, psychiatric, and alcohol and drug use history
* Questions to see if it s safe to have a PET/MRI scan
* Blood and urine tests
* Breath test for alcohol

Participants will have 3 or 4 study visits. At each visit they will have:

* Urine and breath tested for alcohol and drugs
* A thin plastic tube (catheter) inserted in each arm by needle
* A small amount of radioactive chemical injected through the catheter.
* PET/MRI scan. Participants will lie still on a table that slides in and out of a metal cylinder surrounded by a strong magnetic field. Their vital signs will be monitored. They will get earmuffs for loud noises. Before the scan, participants will get the study drug or placebo through the catheter. They may also get a sugar pill (placebo). They will get a small meal and have blood drawn.
* Tests of memory, attention, and thinking.

Participants will wear an activity monitor on the wrist for one week.

DETAILED DESCRIPTION:
Objectives: The overarching goal of this study is to assess the dynamic association between dopamine (DA) D2 receptor (D2R) occupancy measured by positron emission tomography (PET) with [11C]raclopride and brain activity inferred by pharmacological magnetic resonance imaging (phMRI) in the human brain, and to assess the relative sensitivity and specificity of the neurovascular coupling for slow (oral) versus rapid (intravenous, IV) stimulant methylphenidate (MP) delivery. Secondary objectives are to assess the associations between behavioral measures (heart and respiration rates and blood pressure, motor and sleep parameters, and neuropsychological testing variables), D2R occupancy and fMRI signals.

Study population: 10 healthy males and 10 healthy females 18-55 years old will be included. Test-retest reproducibility studies will be carried out in 5 participants.

Design: Double-blind. Participants will undergo simultaneous PET/phMRI, to evaluate dynamic changes in D2R occupancy by DA with [11C]raclopride and in blood-oxygenation-level dependent (BOLD) signals, under MP or placebo (PL). The participants will be scanned on 3 different occasions: 1) oral-MP (60 mg) and iv PL (3 cc saline), 2) oral-PL and iv-MP (0.25 mg/kg in 3 cc sterile water) and 3) oral PL and iv PL, which will be carried in different study days with at least 48 hours between them and their order will be randomized across subjects. Participants and researchers will be blind to the nature of the stimulant drug (MP/PL).

Outcome parameters: The scale factor between the distribution volume ratio (DVR) and the BOLD signal in the dorsal and ventral striatum for the slow and fast MP challenges.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteer Participants

* Males or females between 18 and 55 years of age.
* Ability to provide written informed consent.
* Willing to abstain from drug use on scheduled testing days.
* Have or had any prior experience with alcohol use or stimulant drugs including cocaine, methylphenidate, amphetamine or methamphetamine, diet pills (prescription or over the counter), caffeine, and others but did not have a substance use disorder.

EXCLUSION CRITERIA:

* Pregnant or breastfeeding. Females of childbearing potential must have negative urine pregnancy test and not be currently breastfeeding. Postmenopausal or surgically sterile (tubal ligation or hysterectomy) females satisfy these criteria.
* Unwilling or unable to refrain from use within 24 hours of scheduled study procedures: psychoactive medications or medication that may affect study results (e.g., antibiotics (must finish course at least 24 hours prior to a scheduled procedure), antidiarrheal preparations, anti-inflammatory drugs [systemic corticosteroids are exclusionary], anti-nausea, cough/cold preparations) (self-report, medical history). The following medications are allowable for entry on this study: analgesics (non-narcotic); antacids; antiasthma agents that are not systemic corticosteroids; antifungal agents for topical use; antihistamines (non-sedating); H2-Blockers/proton pump inhibitors (PPI); laxatives. The use of antihyperlipidemics and/or diuretics are permitted if they have been taken for at least 1 month before procedure visits and dose has been stabilized. The episodic use of benzodiazepines such as alprazolam (Xanax), diazepam (Valium) and lorazepam (Ativan), will not exclude participants from this study unless they have been taken within the last 24 hours prior to the study.
* The following current chronically used medications are exclusionary from the study: stimulant or stimulant-like medications (amphetamine, methylphenidate, modafinil); analgesics containing narcotics; anorexics (sibutramine); antianginal agents; antiarrhythmics; antiasthma agents that are systemic corticosteroids; antibiotics; anticholinergics; anticoagulants; anticonvulsants; antidepressants; antidiarrheal preparations; antifungal agents (systemic); antihistamines (sedating); antihypertensives; anti-inflammatory drugs (systemic); antineoplastics; antiobesity; antipsychotics; antivirals (except for treatment of HSV with agents without CNS activity, e.g. acyclovir, ganciclovir, famciclovir, valacyclovir); anxiolytics (benzodiazepine or barbiturates); hormones (exceptions: thyroid hormone replacement, oral contraceptives, and estrogen replacement therapy); insulin; lithium; muscle relaxants; psychotropic drugs not otherwise specified (nos) including herbal products (no drugs with psychomotor effects or with anxiolytics, stimulant, antipsychotic, or sedative properties); sedatives/hypnotics. Note that nicotine and/or caffeine use will not exclude participants.
* Current or past Diagnostic and Statistical Manual (DSM)-IV or DSM-5 diagnosis of a psychiatric disorder as determined by history and clinical exam including substance use disorder (except for nicotine/caffeine), alcohol use disorder (or alcohol dependence, if assessed using DSM-IV) anxiety disorder or panic attacks. Past history of a mental disorder as defined by DSM-IV or DSM-5 will be excluded only if it required hospitalization (any length), or chronic medication management (more than 4 weeks), and that could impact brain function at the time of the study.
* Those with a binge drinking history every month continuously for the last 10 years will also be excluded. Binge drinkers are those who being female consume 4 or more drinks and males consume 5 or more drinks in one occasion at least once a month.
* Major medical problems that can impact brain function at the time of the scan (including but not limited to HIV; glaucoma, central nervous system including seizures and psychosis; cardiovascular including hypertension and arrhythmias; metabolic, autoimmune, endocrine) as determined by history and clinical exam.
* Any clinically significant laboratory finding as determined during the screening procedures.
* Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that, with the exposure from this study, would exceed NIH annual research limits.
* Head trauma with loss of consciousness for more than 30 minutes.
* Presence of ferromagnetic objects in the body that are contraindicated for PET/phMRI of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments), fear of enclosed spaces, or other standard contraindication to MRI/magnetic resonance spectroscopy (MRS) (self-report checklist).
* Cannot lie comfortably flat on back for up to 2 hours in the PET/phMRI scanner.
* Body weight > 204 kg (> 450 lbs).
* Allergy to methylphenidate.
* Clinically significant EKG abnormalities. Clinically significant findings on EKG will be assessed by the Medical Advisory Investigator on the study or through a cardiology consult. EKG reviews are documented in Clinical Research Information System (CRIS).
* History of glaucoma as determined by medical history.
* NIH employees who are study investigators, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).
* Non-English speakers (must also be able to read and comprehend English).

Subjects will not be excluded from enrollment in this study if their urine test is positive for drugs. However, if they test positive on scheduled study procedure days involving study imaging and neuropsychological testing, the procedures will be postponed and rescheduled. We will allow for up to 3 rescheduled study days that were the result of positive urine drug screens. If the drug test is positive on the third rescheduled visit, the participant will be withdrawn from the study. The intent of the research has no prospect of direct benefit to the subject. Therefore, we are excluding non-English speakers in this research study since it includes the administration of questionnaires, surveys and assessments that are validated for English, although some are available in Spanish. In addition,

our fMRI paradigms (particularly the Delay Discounting task) require that the subject be able to speak, read and comprehend English.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dardo G Tomasi, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.Data is analyzed by subject group and not on an individual basis.

REFERENCES:
- [Result] Manza P, Tomasi D, Shokri-Kojori E, Zhang R, Kroll D, Feldman D, McPherson K, Biesecker C, Dennis E, Johnson A, Yuan K, Wang WT, Yonga MV, Wang GJ, Volkow ND. Neural circuit selective for fast but not slow dopamine increases in drug reward. Nat Commun. 2023 Nov 8;14(1):6408. doi: 10.1038/s41467-023-41972-6. PMID 37938560
- [Result] Manza P, Tomasi D, Vines L, Sotelo D, Yonga MV, Wang GJ, Volkow ND. Brain connectivity changes to fast versus slow dopamine increases. Neuropsychopharmacology. 2024 May;49(6):924-932. doi: 10.1038/s41386-024-01803-8. Epub 2024 Feb 7. PMID 38326458
- [Result] Tomasi D, Manza P, Yan W, Shokri-Kojori E, Demiral SB, Yonga MV, McPherson K, Biesecker C, Dennis E, Johnson A, Zhang R, Wang GJ, Volkow ND. Examining the role of dopamine in methylphenidate's effects on resting brain function. Proc Natl Acad Sci U S A. 2023 Dec 26;120(52):e2314596120. doi: 10.1073/pnas.2314596120. Epub 2023 Dec 18. PMID 38109535
- [Result] Tomasi D, Manza P, Logan J, Shokri-Kojori E, Yonga MV, Kroll D, Feldman D, McPherson K, Biesecker C, Dennis E, Johnson A, Yuan K, Wang WT, Butman JA, Wang GJ, Volkow ND. Time-varying SUVr reflects the dynamics of dopamine increases during methylphenidate challenges in humans. Commun Biol. 2023 Feb 10;6(1):166. doi: 10.1038/s42003-023-04545-3. PMID 36765261
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-AA-0178.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants withdrew from the study prior to randomization
Period: Visit Day A (First Intervention)
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo
Started | 8 | 7 | 7
Completed | 8 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Visit Day B (Second Intervention)
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo
Started | 8 | 7 | 7
Randomized to Study Arm A | 0 | 4 | 3
Randomized to Study Arm B | 4 | 0 | 4
Randomized to Study Arm C | 4 | 3 | 0
Completed | 8 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Visit Day C (Third Intervention)
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo
Started | 8 | 7 | 5
Randomized to Study Arm A | 0 | 3 | 4
Randomized to Study Arm B | 4 | 0 | 1
Randomized to Study Arm C | 4 | 4 | 0
Completed | 8 | 7 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Oral Methylphenidate Followed by Intravenous Placebo: Healthy participants receive methylphenidate 60mg orally given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous placebo (3ml saline) given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection.
- Arm B: Oral Placebo Followed by Intravenous Methylphenidate: Healthy participants receive oral placebo given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous methylphenidate 0.25 mg/kg in 3ml sterile water given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection.
- Arm C: Oral Placebo Followed by Intravenous Placebo: Healthy participants receive oral placebo given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous placebo (3ml saline) given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection.
- Total: Total of all reporting groups
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo | Total
Number analyzed (Participants) | 8 | 7 | 7 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 7 | 22
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 7 | 6 | 20
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 3 | 10
  White | 4 | 0 | 3 | 7
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Standardized Uptake Value Ratio (SUVR) for [11C]Raclopride in Putamen
Description: Participants underwent brain positron emission tomography (PET) scan with [11C]raclopride. The SUVR is calculated by dividing the standardized uptake value in the putamen, target region, by the standardized uptake value in the cerebellum, the reference region. This ratio normalizes the uptake values and allows for comparisons between individuals or across different imaging sessions.
Time Frame: 60 min after [11C]raclopride injection
Population: All participants who received [11C]raclopride injection during the PET scans and completed all three arms of the study.
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Groups:
- Arm A: Oral Methylphenidate Followed by Intravenous Placebo Placebo: Healthy participants receive methylphenidate 60mg orally given 30 minutes prior to bolus [11C]raclopride injection followed by intravenous placebo (3ml saline) given 30 minutes post bolus injection of [11C]raclopride. PET/phMRI scan (MRI and PET scan) was initiated at the start of the [11C]raclopride injection. Participants were subsequently randomized across study arms B and C in different study days with at least 48 hours between visits.
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo
Number analyzed (Participants) | 20 | 20 | 20
SUV Ratio (SUVR) | 4.49 (0.39) | 4.39 (0.45) | 4.87 (0.46)

2. Primary Outcome: Percent BOLD Signal Change in the Anterior Cingulum
Description: The blood-oxygen-level-dependent (BOLD) signal was estimated as the fitted amplitude to the dynamic standardized uptake value ratio (SUVR) change in response to the methylphenidate challenges.
Time Frame: From 0 to 90 minutes after [11C]raclopride injection
Population: All participants who received [11C]raclopride injection during the PET scans and completed all three arms of the study.
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo
Number analyzed (Participants) | 20 | 20 | 20
percentage signal change | -0.13 (0.28) | 1.210 (0.620) | -0.001 (0.460)

3. Primary Outcome: The Temporal Correlation Between BOLD(t) and SUVR(t) Change
Description: The Pearson correlation between the temporal dynamics of the blood-oxygen-level-dependent (BOLD) signal in anterior cingulum and the standardized uptake value ratio (SUVR) change in putamen measures changes in the neurovascular coupling induced by methylphenidate.
Time Frame: From 0 to 90 minutes after [11C]raclopride injection
Population: Analysis include all 20 participants who completed the study and received methylphenidate orally and intravenously as pre-specified in the protocol
Measure: Mean (Standard Deviation); unit: correlation coefficient (r)
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate
Number analyzed (Participants) | 20 | 20
correlation coefficient (r) | .023 (.376) | .556 (.219)

ADVERSE EVENTS:
Time Frame: Participants were monitored over 4-6 clinic visits for up to 6 hours per clinic visit
Arm/Group | Arm A: Oral Methylphenidate Followed by Intravenous Placebo | Arm B: Oral Placebo Followed by Intravenous Methylphenidate | Arm C: Oral Placebo Followed by Intravenous Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 10/22 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Oral Methylphenidate Followed by Intravenous Placebo (N=22) | Arm B: Oral Placebo Followed by Intravenous Methylphenidate (N=22) | Arm C: Oral Placebo Followed by Intravenous Placebo (N=22)
Palpitations (Cardiac disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Feeling of relaxation (General disorders) | 1 | 2 | 0
Pain (General disorders) | 0 | 2 | 0
Agitation (Nervous system disorders) | 0 | 3 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Logorrhoea (Nervous system disorders) | 0 | 1 | 0
Restlessness (Nervous system disorders) | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Disturbance in sexual arousal (Psychiatric disorders) | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT03326245/Prot_SAP_000.pdf